CLINICAL TRIAL: NCT06540950
Title: Study of Oral Vinorelbine Single Drug Concurrent Chemoradiotherapy and Immune-maintenance Therapy in Patients With Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Concurrent Chemoradiotherapy With Oral Vinorelbine in Patients With Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3690
Record Dates: First submitted 2024-07-13; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Vinorelbine
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral vinorelbine concurrent radiotherapy group (Experimental): All patients with unresectable stage III non-small cell lung cancer who received neoadjuvant chemo-immunotherapy received oral vinorelbine (60mg per square meter of body-surface area every 2 weeks before radiotherapy, and 30mg per square meter of body-surface area per week during radiotherapy) as radical concurrent chemoratherapy.
  Interventions: Drug: vinorelbine

INTERVENTIONS:
Drug: vinorelbine — Vinorelbine is administered orally at 60mg per square meter per week by body surface area before radiotherapy and continued to be administered at 30mg per square meter per week during radiotherapy until the end of radiotherapy. Within 6 weeks after the end of radiotherapy, there are no serious side effects, and immune checkpoint inhibitors monotherapy can be performed.
  Other Names: oral vinorelbine concurrent chemoradiotherapy

SUMMARY:
To evaluate the efficacy and safety of concurrent chemoradiotherapy with oral vinorelbine, and immune maintenance therapy in patients with unresectable stage III non-small cell lung cancer after neoadjuvant chemo-immunotherapy, with a view to providing an effective treatment regimen for these patients.

DETAILED DESCRIPTION:
Patients with unresectable stage III non-small cell lung cancer after neoadjuvant chemo-immunotherapy are enrolled to receive concurrent chemoradiotherapy with oral vinorelbine, and immune-maintenance therapy. The primary endpoint is objective response rate, and secondary endpoints include disease control rate, progression-free survival, compliance and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years old.
2. Patients must have histologically or cytologically confirmed non-small cell lung cancer.
3. ECOG PS was 0 or 1.
4. Adequate organ and bone marrow function is present. Absolute neutrophil counts, platelet counts, and hemoglobin criteria must not be met after blood transfusion or growth factor support within 14 days prior to randomization.

Exclusion Criteria:

1. History of allogeneic organ transplantation.
2. Active or previously documented autoimmune or inflammatory diseases (including inflammatory bowel disease [Colitis or Crohn's disease], diverticulitis [other than diverticulitis], systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome [granulomatous vasculitis, Graves' disease, rheumatoid arthritis, pituitaritis, uveitis]).
3. There is uncontrolled serious underlying diseases, including active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, uncontrolled arrhythmia, active interstitial lung disease, and severe chronic gastrointestinal disease.
4. History of another primary malignancy.
5. History of active primary immunodeficiency.
6. Histological findings showed mixed small cell lung cancer and non-small cell lung cancer.
7. For any unmitigated toxicity during pre-study chemoradiotherapy. Patients who develop irreversible toxicity and are reasonably expected not to worsen after study treatment (such as hearing loss) may enter the study after consultation with the study physician.
8. Patients who developed ≥ grade 3 pneumonia during study chemoradiotherapy.
9. Received any other concurrent chemotherapy, immunotherapy, biotherapy, or hormonal therapy for cancer other than the therapy evaluated in this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The time between the start of treatment and death from any cause in the one-arm trial
objective response rate | 3 months
  The ratio of complete response and partial response at 3 months after the end of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lei Deng, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lian X, Shayan G, Yang S, Liu W, Zhang T, Lv J, Wang W, Wang J, Wang X, Xiao Z, Zhou Z, Bi N, Deng L. Efficacy and safety of oral vinorelbine with concurrent radiotherapy in unresectable stage III non-small cell lung cancer following neoadjuvant chemoimmunotherapy: a single-arm, phase 2 trial. J Natl Cancer Cent. 2025 Jul 21;5(6):593-599. doi: 10.1016/j.jncc.2025.06.004. eCollection 2025 Dec. PMID 41497257